CLINICAL TRIAL: NCT01721928
Title: Norwegian Intensive Care Unit Dalteparin Effect Study
Acronym: NORIDES
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Sigrid Beitland, Oslo University Hospital, Oslo University Hospital
Other Study IDs: 2012/942; UiO (Other: University of Oslo)
Record Dates: First submitted 2012-10-26; First posted 2012-11-06 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Acute Kidney Injury; Deep Venous Thrombosis
Keywords: Acute kidney injury; Deep venous thrombosis; Dialysis; Prophylaxis
MeSH Terms: conditions — Acute Kidney Injury; Venous Thrombosis | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 12 ml whole blood (10 ml for storage and 2 ml for bedside TEG analysis) will be aspirated from the arterial or the central venous catheter for each measurement. Four measurements will be performed in each patient, from minimum day 2 to maximum day 30 dependent on the dialysis therapy.
  Four urinary samples (each of 20 ml) will be collected from urinary catheter collection bags at the same time as blood samples are drawn.
  Blood (20 mL stored as whole blood, serum and plasma) and urine samples (20 mL) will be collected from each patient at the same time as blood samples are drawn. The samples will be stored at - 70°C for future analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICU patients with AKI: ICU patients with AKI treated with continuous venovenous hemodialysis
  Interventions: Device: Continuous venovenous hemodialysis
- ICU patients without AKI: ICU patients without AKI defined as RIFLE group O and R

INTERVENTIONS:
Device: Continuous venovenous hemodialysis — Continuous venovenous hemodialysis
  Other Names: CVVHD; CRRT
  Groups: ICU patients with AKI

SUMMARY:
The main purpose of the NORIDES study is to investigate the effect of pharmacological thromboprophylaxis with low molecular weight heparins (LMWHs) in critically ill patients, and how it is affected by presence of acute kidney injury (AKI) and treatment with hemodialysis. The main objective is to compare the prophylactic effect of dalteparin in intensive care unit (ICU) patients with AKI and Citrate-Calcium dialysis (CiCa-dialysis) with a control group of ICU patients with normal kidney function. Our main hypothesis is that CiCa-dialysis reduces dalteparin effect, and that patients undergoing CiCa-dialysis do not achieve adequate prophylaxis against venous thromboembolism (VTE). The primary endpoint is development of DVT during ICU stay, the secondary endpoint inadequate heparin effect measured in blood samples.

DETAILED DESCRIPTION:
Description of deep venous thrombosis (DVT) diagnosis: Screening for DVT using Doppler Ultrasound (DUS) of both upper- and lower extremities will be performed within 48 hours after ICU admission and thereafter twice a week until discharge from ICU or ICU stay equal to 30 days. An additional DUS will be performed 3 months after ICU discharge.

Description of heparin effect measured in blood samples: Blood samples will be drawn from intravasal catheters (preferably arterial, alternatively central venous) to examine heparin effect (anti-Xa activity, thrombin generation assay (TGA) and thrombelastography (TEG) and other haematological analyses including antithrombin concentrations. Whole blood will be drawn on two separate days (from minimum day 2 to maximum day 30 dependent on the dialysis therapy) of ICU stay immediately before and 4 hours after dalteparin administration in order to measure tough and peak effect of heparin. Dalteparin effect in ICU patients undergoing dialysis therapy will be measured one day with and one day without ongoing dialysis therapy in order to distinguish the effect of AKI from the effect of continuous renal replacement therapy (CRRT).

ELIGIBILITY:
Inclusion Criteria:

* ICU patients receiving prophylactic dalteparin

Exclusion Criteria:

* Age < 18 years
* Intraocular bleeding
* Intracranial bleeding
* Acute spinal cord lesion
* Inherited coagulopathy
* Ongoing, uncontrolled bleeding
* Therapeutic anticoagulation
* Uncorrected coagulopathy
* Pregnancy or postpartum < 6 weeks
* Participation in an interventional study
* RIFLE class E
* Consent not received
* ICU length of stay less than 48 hours
* DVT detected at first DUS examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The main objective is to compare the prophylactic effect of dalteparin in intensive care unit patients with acute kidney injury and continuous renal replacement therapy with a control group of intensive care unit patients with normal kidney function.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-12-03 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is development of deep venous thrombosis (DVT) | Twice a week until ICU LOS 30 days or discharge from ICU
  Screening for DVT using DUS of both upper- and lower extremities will be performed within 48 hours after ICU admission and thereafter twice a week until discharge from ICU or ICU stay equal to 30 days. An additional DUS will be performed 3 months after ICU discharge.

SECONDARY OUTCOMES:
The secondary endpoint is inadequate heparin effect measured in blood samples | Blood samples is drawn 4 times during ICU stay, from minimum day 2 to maximum day 30 dependent on the dialysis therapy
  Blood samples will be drawn from intravasal catheters (preferably arterial, alternatively central venous) to examine heparin effect (anti-Xa activity, TGA and TEG) and other haematological analyses including antithrombin concentrations. Whole blood will be drawn on two separate days immediately before and 4 hours after dalteparin administration in order to measure tough and peak effect of heparin. Dalteparin effect in ICU patients undergoing dialysis therapy will be measured one day with and one day without ongoing dialysis therapy in order to distinguish the effect of AKI from the effect of CRRT.

OTHER OUTCOMES:
Which of the blood sample analyses anti-Xa activity, TEG or TGA is superior in detecting critically ill patients who will subsequently develop DVT? | Whole blood will be drawn on two separate days from minimum day 2 to maximum day 30 dependent on the dialysis therapy, immediately before and 4 hours after dalteparin administration in order to measure tough and peak effect of heparin.
  The blood sample analyses anti-Xa activity, TEG and TGA will be analysed, and their ability to detect critically ill patients who will subsequently develop DVT. Different patients with and without AKI will be compared. Samples from the same patients one day with and one day without dialysis therapy will also be compared.
Which factors affect heparin effect in critically ill patients? | During ICU stay until LOS 30 days or discharge from ICU
  The following factors will be assessed: Presence of AKI, dialysis therapy, Body mass index (BMI), gender, high severity of illness, use of vasopressors, presence of oedema and serum antithrombin concentrations.
What is the incidence of DVT and bleeding in ICU patients with and without CiCa-dialysis therapy, and is it correlated to heparin effect? | During ICU stay until LOS 30 days or discharge from ICU
  Compare the incidence of DVT and bleeding among ICU patients with and without CiCa-dialysis. Investigate if patient with bleeding have different anti-Xa activity levels, TGA and TEG than patients without bleeding, and if patients with DVT have different anti-Xa activity levels, TGA and TEG compared to patients without DVT.
Do ICU patients with AKI treated with CRRT have lower blood flow to the kidneys measured as renal perfusion index during contrast enhanced DUS compared to similar ICU patients without AKI? | During ICU stay until LOS 30 days or discharge from ICU
  Blood flow to the kidneys measured as renal perfusion index during contrast enhanced DUS will be compared in selected ICU patients with and without CRRT.
Is the renal blood flow measured as renal perfusion index during contrast enhanced DUS correlated to a global blood flow measured as cardiac index using PICCO®? | During ICU stay until LOS 30 days or discharge from ICU
  Blood flow to the kidneys measured as renal perfusion index during contrast enhanced DUS will be compared with global perfusion measured as cardiac index using a pulse contour analysis device (PICCO®).
Is examination of patient urine using Nuclear Magnetic Resonance (NMR) spectroscopy different in ICU patient with and without AKI and what is the effect of CiCa-dialysis on NMR spectroscopy? | During ICU stay until LOS 30 days or discharge from ICU
  NMR spectroscopy of urine in ICU patients with and without AKI necessitating CRRT will be compared, and levels in the same patients with and without dialysis therapy. Further, NMR spectroscopy of urine in the same patient with and without dialysis therapy will be compared.
Which bedside method is superior in predicting dialysis circuit clotting? | During ICU stay until LOS 30 days or discharge from ICU
  Collect data on filter clotting. Evaluate the predictive value of different bedside methods clinically used to forecast filter clotting: Post filter ionised calcium, heparin-active R-time during TEG, access pressure, filter pressure, return pressure and visual inspection of the dialysis circuit air trap.
Which factors affects filter lifetime during CiCa-dialysis? | During ICU stay until LOS 30 days or discharge from ICU
  Collect data on filter lifetime during CiCa-dialysis therapy and investigate if there is a correlation between measured filter lifetime and the following factors: Heparin effect, antithrombin levels, post filter ionised calcium, NMR spectroscopy of urine, clinical assessment of clotting as well as anatomical placement of the dialysis catheter.
Which risk factors for DVT are present in an ICU population and what is the contribution of each factor in development of DVT? | During ICU stay until LOS 30 days or discharge from ICU
  Prospective collection of data on risk factor for DVT in an ICU population according to international guidelines. Also screening for DVT in an ICU population using DUS. Thereafter we plan to perform an analysis on the contribution of each risk factor and combinations of risk factors on development of DVT, with special attention towards possible avoidable risk factors.
Is the presence of DVT in ICU patients influenced by the anatomical placement of catheters such as central venous catheters (CVCs) and dialysis catheters? | During ICU stay until LOS 30 days or discharge from ICU
  Compare the incidence of catheter related DVT if CVC and dialysis catheters are placed in the femoral, subclavian and internal jugular veins.
Does the presence of DVT influence the prognosis in ICU patients? | Data will be collected during ICU stay until LOS 30 days or discharge from ICU. Mortality will also be assessed after ICU discharge.
  To compare preset prognostic markers for morbidity (ICU and hospital length of stay in addition to time on ventilator and dialysis therapy) and mortality (ICU mortality and 30 days mortality) in patients with and without presence of DVT.
Does metabolic alkalosis due to CiCa-dialysis therapy lead to prolonged ventilator therapy? | During ICU stay until LOS 30 days or discharge from ICU
  To compare arterial blood gases in ICU patients with and without CiCa-dialysis and evaluate if patients treated with dialysis more often have metabolic alkalosis. Further, to study whether there is an association between presence of metabolic alkalosis and time spent on ventilator therapy.
What is the compliance to our clinical practice guidelines for thromboprophylaxis in the ICU, and does low compliance to guidelines lead to more frequent DVT? | During ICU stay until LOS 30 days or discharge from ICU
  To compare occurrence of DVT and its correlation to compliance to clinical practice guidelines for DVT prophylaxis, including pharmacological and non-pharmacological prophylaxis.
What is the occurrence of DVT 3 months after ICU discharge? | Patients will be screened for DVT 3 months after ICU discharge.
  To find the occurrence of DVT in critically ill patients 3 months after ICU discharge. Survivors who did not develop DVT during ICU stay will be screened for DVT after 3 months using DUS examination.
Future blood and urine analyses of ICU patients with and without AKI and dialysis therapy. | Blood and urine samples will be collected during ICU stay until LOS 30 days or discharge from ICU. The samples will be stored for future analysis with a maximum of 10 years storage.
  To compare blood and urine samples from critically ill patients with and without AKI and dialysis therapy. The blood and urin samples can be stored for maximum 10 years. The plan is to use new, yet not known analysis methods, and test their utility when assessing ICU patients with and without AKI and dialysis therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Sunde, Professor, Study Chair — Oslo University Hospital; Sigrid Beitland, MD, Principal Investigator — Oslo University Hospital; Per M Sandset, Professor, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Background] McCunn M, Reynolds HN, Reuter J, McQuillan K, McCourt T, Stein D. Continuous renal replacement therapy in patients following traumatic injury. Int J Artif Organs. 2006 Feb;29(2):166-86. doi: 10.1177/039139880602900204. PMID 16552665
- [Background] Cook DJ, Douketis J, Arnold D, Crowther MA. Bleeding and venous thromboembolism in the critically ill with emphasis on patients with renal insufficiency. Curr Opin Pulm Med. 2009 Sep;15(5):455-62. doi: 10.1097/MCP.0b013e32832ea4dd. PMID 19617833
- [Background] Geerts WH, Pineo GF, Heit JA, Bergqvist D, Lassen MR, Colwell CW, Ray JG. Prevention of venous thromboembolism: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):338S-400S. doi: 10.1378/chest.126.3_suppl.338S. PMID 15383478
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271
- [Background] Geerts WH, Heit JA, Clagett GP, Pineo GF, Colwell CW, Anderson FA Jr, Wheeler HB. Prevention of venous thromboembolism. Chest. 2001 Jan;119(1 Suppl):132S-175S. doi: 10.1378/chest.119.1_suppl.132s. No abstract available. PMID 11157647
- [Background] Leclerc JR, Gent M, Hirsh J, Geerts WH, Ginsberg JS. The incidence of symptomatic venous thromboembolism after enoxaparin prophylaxis in lower extremity arthroplasty: a cohort study of 1,984 patients. Canadian Collaborative Group. Chest. 1998 Aug;114(2 Suppl Evidence):115S-118S. doi: 10.1378/chest.114.2_supplement.115s. No abstract available. PMID 9726704
- [Background] Ribic C, Lim W, Cook D, Crowther M. Low-molecular-weight heparin thromboprophylaxis in medical-surgical critically ill patients: a systematic review. J Crit Care. 2009 Jun;24(2):197-205. doi: 10.1016/j.jcrc.2008.11.002. Epub 2009 Feb 7. PMID 19327323
- [Background] Spyropoulos AC, Anderson FA Jr, FitzGerald G, Decousus H, Pini M, Chong BH, Zotz RB, Bergmann JF, Tapson V, Froehlich JB, Monreal M, Merli GJ, Pavanello R, Turpie AGG, Nakamura M, Piovella F, Kakkar AK, Spencer FA; IMPROVE Investigators. Predictive and associative models to identify hospitalized medical patients at risk for VTE. Chest. 2011 Sep;140(3):706-714. doi: 10.1378/chest.10-1944. Epub 2011 Mar 24. PMID 21436241
- [Background] Khouli H, Shapiro J, Pham VP, Arfaei A, Esan O, Jean R, Homel P. Efficacy of deep venous thrombosis prophylaxis in the medical intensive care unit. J Intensive Care Med. 2006 Nov-Dec;21(6):352-8. doi: 10.1177/0885066606292880. PMID 17095499
- [Background] Rabbat CG, Cook DJ, Crowther MA, McDonald E, Clarke F, Meade MO, Lee KA, Cook RJ. Dalteparin thromboprophylaxis for critically ill medical-surgical patients with renal insufficiency. J Crit Care. 2005 Dec;20(4):357-63. doi: 10.1016/j.jcrc.2005.09.009. PMID 16310608
- [Background] Crowther MA, Cook DJ, Griffith LE, Devereaux PJ, Rabbat CC, Clarke FJ, Hoad N, McDonald E, Meade MO, Guyatt GH, Geerts WH, Wells PS. Deep venous thrombosis: clinically silent in the intensive care unit. J Crit Care. 2005 Dec;20(4):334-40. doi: 10.1016/j.jcrc.2005.09.011. PMID 16310604
- [Background] Douketis JD, Rabbat C, Crowther MA; VTE in the ICU Workshop Participants. Anticoagulant prophylaxis in special populations with an indwelling epidural catheter or renal insufficiency. J Crit Care. 2005 Dec;20(4):324-9. doi: 10.1016/j.jcrc.2005.09.001. PMID 16310603
- [Background] Cook D, Crowther MA, Douketis J; VTE in the ICU Workshop Participants. Thromboprophylaxis in medical-surgical intensive care unit patients. J Crit Care. 2005 Dec;20(4):320-3. doi: 10.1016/j.jcrc.2005.09.007. No abstract available. PMID 16310602
- [Background] Cook D, Douketis J, Crowther MA, Anderson DR; VTE in the ICU Workshop Participants. The diagnosis of deep venous thrombosis and pulmonary embolism in medical-surgical intensive care unit patients. J Crit Care. 2005 Dec;20(4):314-9. doi: 10.1016/j.jcrc.2005.09.003. No abstract available. PMID 16310601
- [Background] Cook DJ, Crowther MA, Meade MO, Douketis J; VTE in the ICU Workshop Participants. Prevalence, incidence, and risk factors for venous thromboembolism in medical-surgical intensive care unit patients. J Crit Care. 2005 Dec;20(4):309-13. doi: 10.1016/j.jcrc.2005.09.005. No abstract available. PMID 16310600
- [Background] Cook DJ, Crowther MA, Geerts WH. On the need for a workshop on venous thromboembolism in critical care. J Crit Care. 2005 Dec;20(4):306-8. doi: 10.1016/j.jcrc.2005.09.004. No abstract available. PMID 16310599
- [Background] Swarczinski C, Dijkers M. The value of serial leg measurements for monitoring deep vein thrombosis in spinal cord injury. J Neurosci Nurs. 1991 Oct;23(5):306-14. doi: 10.1097/01376517-199110000-00007. PMID 1835995
- [Background] Makris PE, Pithara E. Clinical evaluation of new global clotting assay for monitoring of LMWH treatment: pilot study. Int Angiol. 1998 Jun;17(2):69-79. PMID 9754892
- [Background] Haas FJ, Kluft C, Biesma DH, Schutgens RE. Patients with deep venous thrombosis and thrombophilia risk factors have a specific prolongation of the lag time in a chromogenic thrombin generation assay. Blood Coagul Fibrinolysis. 2011 Sep;22(6):506-11. doi: 10.1097/MBC.0b013e328347404d. PMID 21537160
- [Background] Marik PE, Andrews L, Maini B. The incidence of deep venous thrombosis in ICU patients. Chest. 1997 Mar;111(3):661-4. doi: 10.1378/chest.111.3.661. PMID 9118705
- [Background] Cook DJ, Rocker G, Meade M, Guyatt G, Geerts W, Anderson D, Skrobik Y, Hebert P, Albert M, Cooper J, Bates S, Caco C, Finfer S, Fowler R, Freitag A, Granton J, Jones G, Langevin S, Mehta S, Pagliarello G, Poirier G, Rabbat C, Schiff D, Griffith L, Crowther M; PROTECT Investigators; Canadian Critical Care Trials Group. Prophylaxis of Thromboembolism in Critical Care (PROTECT) Trial: a pilot study. J Crit Care. 2005 Dec;20(4):364-72. doi: 10.1016/j.jcrc.2005.09.010. PMID 16310609
- [Background] Patel R, Cook DJ, Meade MO, Griffith LE, Mehta G, Rocker GM, Marshall JC, Hodder R, Martin CM, Heyland DK, Peters S, Muscedere J, Soth M, Campbell N, Guyatt GH; Burden of Illness in venous ThromboEmbolism in Critical care (BITEC) Study Investigators; Canadian Critical Care Trials Group. Burden of illness in venous thromboembolism in critical care: a multicenter observational study. J Crit Care. 2005 Dec;20(4):341-7. doi: 10.1016/j.jcrc.2005.09.014. PMID 16310605
- [Background] Crowther MA, Cook DJ, Griffith LE, Meade M, Hanna S, Rabbat C, Bates SM, Geerts W, Johnston M, Guyatt G. Neither baseline tests of molecular hypercoagulability nor D-dimer levels predict deep venous thrombosis in critically ill medical-surgical patients. Intensive Care Med. 2005 Jan;31(1):48-55. doi: 10.1007/s00134-004-2467-2. Epub 2004 Dec 9. PMID 15592816
- [Background] Cook D, Meade M, Guyatt G, Griffith L, Granton J, Geerts W, Crowther M; Canadian Critical Care Trials Group. Clinically important deep vein thrombosis in the intensive care unit: a survey of intensivists. Crit Care. 2004 Jun;8(3):R145-52. doi: 10.1186/cc2859. Epub 2004 May 6. PMID 15153243
- [Background] Malinoski D, Jafari F, Ewing T, Ardary C, Conniff H, Baje M, Kong A, Lekawa ME, Dolich MO, Cinat ME, Barrios C, Hoyt DB. Standard prophylactic enoxaparin dosing leads to inadequate anti-Xa levels and increased deep venous thrombosis rates in critically ill trauma and surgical patients. J Trauma. 2010 Apr;68(4):874-80. doi: 10.1097/TA.0b013e3181d32271. PMID 20386282
- [Background] Malinoski D, Ewing T, Patel MS, Jafari F, Sloane B, Nguyen B, Barrios C, Kong A, Cinat M, Dolich M, Lekawa M, Hoyt DB. Risk factors for venous thromboembolism in critically ill trauma patients who cannot receive chemical prophylaxis. Injury. 2013 Jan;44(1):80-5. doi: 10.1016/j.injury.2011.10.006. Epub 2011 Nov 1. PMID 22047757
- [Background] Van PY, Cho SD, Underwood SJ, Morris MS, Watters JM, Schreiber MA. Thrombelastography versus AntiFactor Xa levels in the assessment of prophylactic-dose enoxaparin in critically ill patients. J Trauma. 2009 Jun;66(6):1509-15; discussion 1515-7. doi: 10.1097/TA.0b013e3181a51e33. PMID 19509608
- [Background] Klein SM, Slaughter TF, Vail PT, Ginsberg B, El-Moalem HE, Alexander R, D'Ercole F, Greengrass RA, Perumal TT, Welsby I, Gan TJ. Thromboelastography as a perioperative measure of anticoagulation resulting from low molecular weight heparin: a comparison with anti-Xa concentrations. Anesth Analg. 2000 Nov;91(5):1091-5. doi: 10.1097/00000539-200011000-00009. PMID 11049889
- [Background] Schleyer AM, Schreuder AB, Jarman KM, Logerfo JP, Goss JR. Adherence to guideline-directed venous thromboembolism prophylaxis among medical and surgical inpatients at 33 academic medical centers in the United States. Am J Med Qual. 2011 May-Jun;26(3):174-80. doi: 10.1177/1062860610382289. Epub 2011 Apr 13. PMID 21490270